CLINICAL TRIAL: NCT06751758
Title: Effects of Sub Occipital Distraction Versus Manual Traction on Upper Cervical Pain, Range of Motion and Functional Disability in Chronic Neck Pain
Brief Title: Suboccipital Distraction vs. Manual Traction in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Noor Fatima
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cervical Pain
Keywords: Cervical pain; Suboccipital Distraction; Manual Traction; Functional disability; Range of motion
MeSH Terms: conditions — Neck Pain | interventions — Transcutaneous Electric Nerve Stimulation; Traction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Suboccipital Distraction (Experimental): In addition to the initial conservative treatment phase (cervical spine mobilization targeting the C1-C2 region and a 20-minute session of Transcutaneous Electrical Nerve Stimulation (TENS)), participants in Group A will undergo suboccipital distraction as part of the subsequent intervention. Suboccipital distraction involves the gentle separation of the suboccipital muscles and associated structures to alleviate tension and promote relaxation. This technique specifically targets upper cervical pain and aims to enhance range of motion.
  Interventions: Other: C1-C2 Mobilization; Other: Transcutaneous Electrical Nerve Stimulation (TENS); Other: Suboccipital Distraction
- Group B - Traction (Active Comparator): After the initial conservative treatment phase (cervical spine mobilization targeting the C1-C2 region and a 20-minute session of Transcutaneous Electrical Nerve Stimulation (TENS)), participants in Group B will receive traction as their intervention. Traction involves the application of controlled force to stretch and mobilize the cervical spine manually. The aim is to reduce compression on cervical structures, alleviate pain, and improve the range of motion.
  Interventions: Other: C1-C2 Mobilization; Other: Transcutaneous Electrical Nerve Stimulation (TENS); Other: Traction

INTERVENTIONS:
Other: C1-C2 Mobilization — Participants in both Group A and Group B will receive manual mobilization targeting the C1-C2 region. This specific mobilization technique is chosen for its potential to improve joint mobility and alleviate stiffness in the upper cervical spine. The mobilization will be performed by trained physiotherapists to ensure precision and safety.
Other: Transcutaneous Electrical Nerve Stimulation (TENS) — Following C1-C2 mobilization, each participant will undergo a 20-minute session of TENS. TENS involves the application of low-voltage electrical currents through electrodes placed on the skin. This modality aims to modulate pain perception by stimulating nerve fibers, leading to the release of endorphins - the body's natural painkillers. The 20-minute duration is chosen based on established guidelines for effective TENS application.
Other: Suboccipital Distraction — Suboccipital distraction is a manual technique aimed at relieving tension in the upper cervical spine. This intervention involves the gentle separation of the suboccipital muscles and associated structures, promoting relaxation and reducing pain. The technique is intended to enhance the range of motion in the cervical region by targeting the upper cervical structures.
  Procedure:
  5-7 repetitions of intermittent distraction 20-30 seconds on, 10-15 seconds off
  Administration:
  Suboccipital distraction will be performed by skilled physiotherapists trained in this technique. Close monitoring will ensure correct application and participant safety.
  Arms: Group A - Suboccipital Distraction
Other: Traction — Traction is a therapeutic technique that involves applying a controlled, manual force to stretch and mobilize the cervical spine. The primary goal of this intervention is to reduce compression on the cervical structures, alleviate pain, and improve the range of motion. It is typically used for its potential to decompress the spine and relieve pressure on nerves.
  Procedure:
  Traction will be administered manually by trained physiotherapists, who will ensure that the correct amount of force is applied and that the treatment is both safe and effective. The application will be carefully tailored to the individual's needs.
  Administration:
  Participants will undergo traction treatments with close monitoring throughout the study period, allowing for necessary adjustments to the treatment plan based on individual responses.
  Arms: Group B - Traction

SUMMARY:
This study addresses the pervasive issue of chronic neck pain, a debilitating condition with profound implications for daily life and well-being. Two therapeutic techniques, suboccipital distraction, and manual traction, are under investigation for their potential to alleviate upper cervical pain and enhance mobility in individuals suffering from chronic neck pain. The primary goal is to compare the effects of these interventions on upper cervical pain, range of motion, and functional disability, providing valuable insights for healthcare professionals to optimize treatment strategies and enhance outcomes in this challenging context. The research adopts a Randomized Clinical Trial (RCT) design to rigorously evaluate the impact of suboccipital distraction and manual traction on upper cervical pain, range of motion, and functional disability in chronic neck pain patients. The Gpower t-test sample size calculation ensures a robust sample size, enhancing statistical power and the validity of findings. Participants will be recruited from Neuro clinic, Lahore, using non-probability convenient sampling. The lottery method will be employed for randomizing participants into suboccipital distraction and manual traction groups, ensuring a balanced distribution of key characteristics. The diverse patient population at Neuro Clinic enhances the generalizability of the study's results. The treatment plan spans 4 weeks, comprising three sessions per week. Each session involves three sets of suboccipital distraction or manual traction, with 5 to 7 repetitions per set. Baseline assessments will be conducted, followed by post-treatment assessments at the 4-week mark. Outcome measures, including standardized pain scales, goniometry for range of motion, and validated instruments for functional disability, will be systematically collected during these intervals.

DETAILED DESCRIPTION:
Chronic neck pain is a prevalent and debilitating condition affecting a substantial portion of the global population (1). Among the various therapeutic interventions, suboccipital distraction and manual traction emerge as two distinctive approaches, each holding promise in alleviating upper cervical pain, improving range of motion, and enhancing functional disability (2). The upper cervical region, comprising the atlas and axis vertebrae, plays a crucial role in supporting the head's weight and facilitating complex movements (3). Dysfunction in this area can lead to persistent pain and restricted mobility, warranting effective interventions for improved patient outcomes. This study aims to delve into the comparative effectiveness of suboccipital distraction versus manual traction, exploring their impact on upper cervical pain, range of motion, and functional disability in individuals suffering from chronic neck pain. Chronic neck pain is a multifaceted issue, often stemming from a combination of structural, biomechanical, and psychosocial factors (4). The upper cervical spine is particularly susceptible to dysfunction due to its intricate anatomy and constant engagement in supporting the head's movements. Suboccipital distraction, involving the gentle separation of the atlas and axis vertebrae, has gained attention as a therapeutic technique that targets specific structures in the upper cervical region. On the other hand, manual traction, characterized by the application of force to elongate the cervical spine, is another widely used intervention. Despite the prevalence of these approaches, there is a paucity of research directly comparing their efficacy in the context of chronic neck pain. Understanding the nuanced effects of suboccipital distraction and manual traction is crucial for optimizing treatment strategies and tailoring interventions to individual patient needs. Chronic neck pain is a multifaceted issue that affects a significant portion of the global population, with variations in prevalence across different regions. Studies conducted in Asia have reported a considerable number of individuals suffering from chronic neck pain. For instance, a survey in Japan found that approximately 23% of the population experienced persistent neck pain (5). In Europe, studies indicate varying prevalence rates, with a cross-European investigation estimating the prevalence to be around 15% (6). The situation in North America is also noteworthy, with a study conducted in the United States revealing that about 20% of the adult population reported chronic neck pain lasting more than three months (7). These regional disparities highlight the need for comprehensive research that considers diverse populations. Understanding the prevalence of chronic neck pain in different continents is crucial for contextualizing the importance of interventions such as suboccipital distraction and manual traction. Rationale for this study lies in the need for evidence-based guidance in selecting the most effective intervention for chronic neck pain, especially focusing on the upper cervical region. By comparing the outcomes of suboccipital distraction and manual traction, this research aims to contribute valuable insights into their respective impacts on pain reduction, range of motion improvement, and functional disability alleviation. Such knowledge is essential for clinicians seeking to provide personalized and efficient care to patients grappling with chronic neck pain. Moreover, the comparative effectiveness of these interventions can inform future treatment protocols, guiding healthcare professionals in making informed decisions based on empirical evidence. As the burden of chronic neck pain continues to rise globally, optimizing therapeutic approaches becomes imperative, and this study strives to bridge existing gaps in knowledge, paving the way for more effective and targeted interventions. The significance of this study is underscored by the potential implications for clinical practice and patient outcomes. With chronic neck pain being a widespread and often persistent condition, identifying the most effective intervention can substantially improve the quality of life for affected individuals. Suboccipital distraction and manual traction represent distinct therapeutic modalities, and a direct comparison will offer valuable insights into their relative efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Minimum chronicity: of 3 months chronic neck pain (21)
* Spurling test (22)

Exclusion Criteria:

* Chronic systemic bony diseases
* Degenerative joint diseases
* Psychiatric diseases
* Recent history of trauma

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS (Numerical Pain Rating Scale) | baseline, after 4 weeks
  The NPRS is a self-report measure used to assess the intensity of pain experienced by individuals. Participants rate their pain on a numerical scale from 0 (no pain) to 10 (worst possible pain). It is known for its simplicity and ease of administration, making it a practical tool in clinical and research settings.
  Psychometric Properties:
  Validity: Strong convergent validity demonstrated in studies such as Jensen et al. (1986), which compared NPRS with other established pain measures.
  Reliability: The NPRS has been shown to have good test-retest reliability, with consistent pain ratings over time.
  Usefulness: Widely used in clinical settings due to its solid psychometric properties, making it valuable for assessing pain intensity in various populations.
Goniometer | baseline, after 4 weeks
  The goniometer is a fundamental tool for objectively measuring joint range of motion (ROM). It consists of a protractor-like device that quantifies the angular displacement of a joint during movement. Validity and reliability of goniometric measurements are crucial to ensure accurate and consistent assessments. Previous research, such as the work by Norkin and White (2009), has supported the concurrent validity of goniometry by comparing its measurements with those obtained through radiographic imaging (25). The goniometer's well-established validity and reliability make it an indispensable tool for assessing joint mobility and tracking changes in range of motion over time.
NDI | baseline, after 4 weeks
  This will be used to measure function of neck.Neck disability index was the first tool to measure the self-reported disability in patients with neck pain. It has significant psychometric features and has been shown to be very responsible in clinical trials.
  The index has 10 neck-related functional activities scored on a 0-5 likert scale for each item and total score of 50. Higher score on the scale shows greater disability.
  The NDI has very good reliability (ICC = 0.88;[0.63 to 0.95]) (26, 27).

CONTACTS AND LOCATIONS:
Overall Officials: Noor Fatima, DPT, Principal Investigator — Riphah International University, Lahore
Locations (1):
- Neuro Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No